CLINICAL TRIAL: NCT03634202
Title: Phase-1 Study of Escalated-dose Pelvic Radiation Therapy Using Intensity-Modulated Radiotherapy (IMRT) With Simultaneous Integrated Boost (SIB), in Combination With Xeloda, for Initially Metastatic, Low and Middle Rectal Cancer
Brief Title: Study of Radiation Therapy in Combination With Xeloda, for Initially Metastatic, Low and Middle Rectal Cancer
Acronym: DESIR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the study was stopped for lack of inclusion
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICO-A-2013-06
Record Dates: First submitted 2018-08-06; First posted 2018-08-16 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Rectal Cancer; Metastasis; Radiotherapy
Keywords: Intensity Modulated Radiotherapy; Simultaneous Integrated Boost; Low and middle Rectal carcinoma
MeSH Terms: conditions — Rectal Neoplasms; Neoplasm Metastasis | interventions — Radiotherapy, Intensity-Modulated; Drug Therapy; Capecitabine

STUDY DESIGN:
Intervention Model Description: Phase-1 study of escalade dose of radiation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMRT + oral chemotherapy (Experimental): Radiotherapy = IMRT with SIB. The overall duration of irradiation is 5 to 7 weeks Chemotherapy = oral capecitabine. Chemotherapy is taken in concomitance as radiotherapy days
  Interventions: Combination Product: IMRT + oral chemotherapy

INTERVENTIONS:
Combination Product: IMRT + oral chemotherapy — It's a dose escalation of radiation (IMRT), during 5 to 7 weeks, 5 days per week.
  Concomitantly, patient have oral chemotherapy (capecitabin)
  Other Names: Intensity-Modulated Radiotherapy + capecitabine

SUMMARY:
In initially metastatic rectal carcinoma, a neo-adjuvant multi-drug chemotherapy is usually performed, followed by a pelvic chemoradiation. The surgical indications on both metastases and the pelvic site are then discussed: in the case where a complete (or near-complete) response (CR) of the rectal tumor is observed (10 to 40%), the local surgery may be omitted or poned ("wait-and-see") in a sphincter-sparing strategy, in order to minimize or avoid the surgical morbidity, to focus on metastatic disease by the continuation of chemotherapy, and to preserve a better quality of life. After 8 weeks of induction chemotherapy (mFolfox6 regimen, 4 cycles), the aim of our study is to optimize the chemoradiation step on the distal rectal tumor, thanks to Intensity-Modulated Radiotherapy (IMRT) with simultaneous integrated boost (SIB) (Phase-1 part of the study), concomitantly with oral capecitabine. According to a Fibonacci dose-escalation scheme, 3 radiation dose-levels are defined, up to the definition of the maximal tolerated dose (MTD), requiring the inclusion of a maximum of 20 patients. Further patients will be included at the recommended dose for phase-2 (RDP2) in a two-step phase-2 study, considering simultaneously as principal objective at 12 months, both the efficacy (local CR rate in the range of 10 to 25%) and the tolerance (pelvic radiation disease: grade 3-4 toxicities in the range of 30 to 10%). Overall 65 patients will be included in the phase-2 study at the RDP2 dose.

DETAILED DESCRIPTION:
The study population has metastatic rectal cancer. After obtaining informed consent and if they fulfil all of the criteria for inclusion, patients will be included.

After 8 weeks of induction chemotherapy with FOLFOX, patients perform an imaging assessment.

Then they are treated by radiotherapy with an oral Xeloda At the end of irradiation, patients realize on other Imaging assessment. Patients are then followed for 2 years

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic distal rectal carcinoma (low and middle);
2. age >18 years
3. Estimated life expectancy greater than 3 months
4. PS: ECOG<2
5. Normal hematologic, renal and hepatic functions
6. Normal or only partially decreased DPD activity
7. Effective contraception in women and men of childbearing age
8. Social insurance.
9. Signed informed consent

Exclusion Criteria:

1. No previous treatment with pelvic radiotherapy or chemotherapy
2. Disorder precluding understanding of trial information or informed consent
3. No severe or uncontrolled disease (infection, VIH, HBs, diabetes mellitus)
4. No peripheral neuropathy > grade 2
5. No inflammatory disease or fructosemia
6. Diarrhea of grade > 2
7. Pregnancy, breastfeeding women
8. Patients already included in another therapeutic within a period of 30 days
9. Other malignancy treated within the last 5 years (except non-melanoma skin cancer)
10. Bilateral total hip prosthesis
11. Patient is willing and able to comply with the protocol for the duration of the study including all scheduled treatment, visits and examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
maximum tolerated radiation dose (MTD) delivered by IMRT with SIB, in combination with oral capecitabine, for initially metastatic, low and middle rectal cancer after 4 induction cycles of mFolfox6 regimen. | 84 months
  MTD = dose level -1 after at least 2 patients with DLT to upper level

SECONDARY OUTCOMES:
Local Progression-free survival at 12 months, | 12 months after inclusion
  % patient with Local Progression at CT scan, 12 months after inclusion
Toxicity profile of the chemoradiation step for NCI.CTC grade 3-4 local toxicities due to "Pelvic Radiation Disease" | 84 months
  % patient with >= grade 3 toxicity (NCI.CTC AE)
To evaluate quality of Life | 84 months
  EORTC-QLQC-30
To evaluate quality of Life | 84 months
  QLQ-CR29
Overall survival at 2 years | 24 months after inclusion
  Overall survival is defined as the delay between the date of inclusion and the date of end of study
The usefulness of surgery | 12 months after the end of radiochemotherapy
  The surgical decision within 12 months after the end of radiochemotherapy will be recovered
The prognostic value of PET | 108 months
  The interest of PET to define the volume in radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: AMAURY PAUMIER, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- Institut de Cancérologie de l'Ouest, Angers, France

IPD SHARING:
Plan to Share IPD: No